CLINICAL TRIAL: NCT05925257
Title: Design and Evaluation of the Effectiveness of a Digital Health Intervention to Improve Health Care and Outcomes for Cancer Patients
Brief Title: Digital Health Intervention to Improve Health Care and Outcomes for Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Svetlana Doubova, Head of the Epidemiology and Health Services Research Unit National Medical Center Century XXI of the Mexican Institute of Social Security and Principal Investigator of the present study, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R-2021-785-059
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Nurses

STUDY DESIGN:
Intervention Model Description: unblinded, parallel-arm randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be given access to the ePRO application and proactive clinical care, including study nurses responding to ePROs and weekly health information videos for six months.
  Interventions: Other: ePRO application and proactive clinical care with nurses.
- Control group (No Intervention): Participants of the control group will be provided with a list of electronic links to videos on breast cancer-relevant topics on the websites of recognised cancer associations and health institutions.

INTERVENTIONS:
Other: ePRO application and proactive clinical care with nurses. — The investigators defined ePRO intervention as a weekly register of breast cancer patients' symptoms and supportive care needs using the study ePRO App combined with proactive follow-up by nurses guided by predefined clinical algorithms and a weekly cellphone message providing an educational video from a recognised cancer association or health institution. The intervention will be provided for six months with additional three months of post-intervention observation.
  Arms: Intervention group

SUMMARY:
Background: Nearly 30,000 Mexican women develop breast cancer annually. These patients frequently present multiple unmet supportive care needs. In high-income settings, incorporating electronic patient-reported outcomes (ePROs) into cancer care has demonstrated potential for increasing patient-centred care and reducing unmet needs. No such ePRO interventions have been implemented in Mexico. The objectives of this study are (I) to design a two-component intervention for monitoring ePROs among breast cancer patients using a responsive digital application and proactive follow-up by nurses, (II) to perform intervention pilot testing of the study materials, and (III) to conduct the clinical trial to assess usability and effectiveness of the intervention.

Methods. The investigators designed a two-component intervention for women receiving breast cancer treatment: a responsive web application for monitoring ePROs and clinical algorithms guiding proactive follow-up by nurses. The investigators will conduct a pilot test of the intervention with 50 breast cancer patients for six weeks to assess the feasibility and inform intervention adaptations. After that, the investigators will conduct a parallel arm randomized controlled trial assigning 205 patients each to intervention and control in one of Mexico's largest public oncology hospitals. The intervention will be provided for six months, with additional three months of post-intervention observation. The control group will receive usual healthcare and a list of information sources on relevant breast cancer topics. Women diagnosed with stages I, II, or III breast cancer who initiate chemo and/or radiotherapy will be invited to participate. The study outcomes will include supportive care needs, quality of life, use of emergency services and unscheduled hospitalizations, the usability of the ePRO App, and adherence to the intervention. Information on the outcomes will be obtained through web-based self-administered questionnaires collected at baseline, 1, 3, 6, and 9 months.

DETAILED DESCRIPTION:
An unblinded, parallel-arm, randomized, controlled clinical trial will be conducted. This phase 2 clinical trial focuses on exploring the effect of the intervention on the study variables.The intervention group will be given access to the ePRO application and proactive clinical care, including study nurses responding to ePROs and weekly health information videos for six months. Participants of the control group will be provided with a list of electronic links to videos on breast cancer-relevant topics on the websites of recognised cancer associations and health institutions. All participants will continue to receive the usual health care provided by the hospital. Study intervention wil last 6 months with additional passive folow-up till 9 months to allow post-intervention monitoring.

The participants will be randomly allocated to the intervention or control groups. The minimization technique with MS-DOS Minim program will be used for randomization. It will be conducted by a research assistant who will use a pre-prepared list of random numbers to randomize the first six participants. Starting with the seventh participant, randomization will be carried out using MS-DOS Minim program. The minimization technique is recommended as a standard to ensure that clinical trial groups are similar in terms of participant characteristics, such as age, schooling, breast cancer stage and treatment modality.

Intervention implementation: The lead researcher will weekly obtain the list of breast cancer patients who have started or will start neoadjuvant or adjuvant treatment with chemotherapy or radiotherapy within two weeks in the oncology hospital. The previously trained nurses will use this list to invite all eligible breast cancer patients to participate in the study. Initially, patients will be invited by telephone calls to attend the hospital or the research unit (located at the same medical center as the oncology hospital) to receive the study-related information and to confirm eligibility. Those who meet the inclusion criteria will be provided with the option to participate and invited to provide informed consent prior to participation. Participants will be provided with a username, password, and access to the intervention or control interface of the responsive ePRO App, and training on its use. All participants will be asked to answer the baseline record of sociodemographic and clinical characteristics and questionnaires to assess study outcomes. Intervention arm participants will be asked to complete the weekly register and will receive weekly WhatsApp reminders. Study nurses will contact patients without two weekly records to encourage adherence to the intervention. Study nurses will be supported by the study oncologist/ oncology resident to ensure adherence to the intervention activities. Additionally, the nurses will be in regular contact with the study team and will record their activities in the corresponding interface of the responsive ePRO App.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age between 20 and 75 years
* Breast cancer stages I, II, or III
* Neoadjuvant or adjuvant treatment with chemotherapy that started within two to six weeks before enrollment
* Access to the internet on mobile phone, computer or tablet
* Written informed consent

Exclusion Criteria:

* Illiterate
* Stage IV breast cancer
* Cognitive dysfunction
* Blindness or low vision not corrected with glasses
* Severe depression (≥12 points on the Hospital Anxiety and Depression Scale)

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Health systems and information supportive care needs | At 1, 3, 6 and 9 months after intervention commencement
  Change from baseline in health systems and information supportive care needs at 1, 3, 6 and 9 months after the intervention commencement, which will be measured with the Supportive Care Needs Survey Short Form-34 (SCNS SF-34) questionnaire validated in Mexico.

SECONDARY OUTCOMES:
Global quality of life | At 1, 3, 6 and 9 months after intervention commencement
  Change from baseline in Global quality of life at 1, 3, 6 and 9 months after the intervention commencement, which will be measured with the EORTC (European Organization for Research and Treatment of Cancer) QLQ-C30 questionnaire validated in Mexico
Breast symptoms | At 1, 3, 6 and 9 months after intervention commencement
  Change from baseline in breast symptoms at 1, 3, 6 and 9 months after the intervention commencement, which will be measured with the breast symptoms scale of the EORTC QLQ-BR23 questionnaire validated in Mexico.

OTHER OUTCOMES:
Use of emergency services | At 1, 3, 6 and 9 months after intervention commencement
  Change from baseline in the emergency room visits, which will be measured by the number of the emergency room visits during the previous month
Use of the responsive ePRO App in the intervention group | At 1, 3 and 6 months after intervention commencement
  Frequency of the responsive ePRO App use (site visits by IP address) and completion of a weekly report of symptoms and supportive care needs on the responsive digital App.
Unscheduled hospitalizations | At 1, 3, 6 and 9 months after intervention commencement
  Change from baseline in the unscheduled hospitalizations, which will be measured by the number of unscheduled hospitalizations in the previous month
Perceived usability of the responsive ePRO App in the intervention group | At 1, 3 and 6 months after intervention commencement
  Perceived usability will be measured by mHealth Application Usability Questionnaire [ ] translated into Spanish with content validation completed by the study expert group.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana V. Doubova, MD. DSc., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (3):
- Mexico (3):
  - Hospital de Oncología del Centro Médico Nacional Siglo XXI, Mexico City, Mexico City
  - UMAE Hospital de Gineco-Obstetricia No.3 "Dr. Víctor Manuel Espinoza de los Reyes Sánchez" CMN La Raza., Mexico City
  - UMAE Hospital de Especialidades CMN "Gral. de Div. Manuel Ávila Camacho", Puebla City

IPD SHARING:
Plan to Share IPD: Yes
De-identified study variables will be available.
Supporting Information: Study Protocol
Time Frame: De-identified data will be available once a trial is completed and their primary results are published and for 5 years thereafter.
Access Criteria: De-identified study variables will be available to secondary researchers whose proposed research has received IRB approval.

REFERENCES:
- [Derived] Contreras Sanchez SE, Doubova SV, Martinez Vega IP, Grajales Alvarez R, Villalobos Valencia R, Dip Borunda AK, Lio Mondragon L, Martinez Pineda WJ, Nunez Cerrillo JG, Huerta Lopez AD, Zalapa Velazquez R, Mendoza Ortiz V, Vazquez Zamora VJ, Montiel Jarquin AJ, Garcia Galicia A, Talamantes Gomez EI, Sanchez Reyes R, Aguirre Gomez J, Ayala Anzures ME, Zapata Tarres M, Monroy A, Leslie HH. Addressing the unmet needs of women with breast cancer in Mexico: a non-randomised pilot study of the digital ePRO intervention. BMJ Open. 2024 Jun 21;14(6):e087240. doi: 10.1136/bmjopen-2024-087240. PMID 38908841
- [Derived] Contreras Sanchez SE, Doubova SV, Grajales Alvarez R, Dip Borunda AK, Martinez Pineda WJ, Nunez Cerrillo JG, Silva Bravo F, Zalapa Velazquez R, Gutierrez De la Barrera M, Leslie HH. Design and evaluation of a digital health intervention with proactive follow-up by nurses to improve healthcare and outcomes for patients with breast cancer in Mexico: protocol for a randomised clinical trial. BMJ Open. 2023 Nov 6;13(11):e077322. doi: 10.1136/bmjopen-2023-077322. PMID 37931967